CLINICAL TRIAL: NCT00601055
Title: Treating Older Patients With Major Depression and Severe COPD
Brief Title: Problem-Solving Therapy for People With Major Depression and Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH076829 (NIH); 0511008253 (Other: Weill Cornell IRB Protocol Number); R01MH076829 (NIH); NCT00504569 (obsolete NCT alias)
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Depression
Keywords: COPD; Geriatric Depression; Problem-Solving Therapy; Treatment Adherence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Depression; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Problem Solving-Rx Adherence (PSA) (Experimental): Participants will receive problem-solving therapy integrated with adherence-enhanced procedures (PSA).
  Interventions: Behavioral: Problem Solving-Rx Adherence (PSA)
- PID-C (Active Comparator): Participants will receive adherence-enhanced (PID-C) procedures, a treatment mobilizing patients to participate in their care.
  Interventions: Behavioral: PID-C

INTERVENTIONS:
Behavioral: Problem Solving-Rx Adherence (PSA) — In PSA, a therapist teaches the participant to identify problems related to depression, functioning, and treatment adherence; to generate multiple solutions; and to choose and implement one or more of those solutions.
  Arms: Problem Solving-Rx Adherence (PSA)
Behavioral: PID-C — In PID-C, a therapist identifies obstacles to treatment adherence and helps the participant overcome those obstacles.
  Arms: PID-C

SUMMARY:
This study will evaluate the effectiveness of problem-solving therapy combined with treatment adherence procedures in treating older people with major depression and chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Depression is a serious illness that affects a person's mood, thoughts, and physical well-being. Common symptoms of depression include persistent feelings of anxiety, guilt, or hopelessness; irregular sleep and appetite patterns; lethargy; disinterest in previously enjoyed activities; excessive irritability and restlessness; suicidal thoughts; and inability to concentrate. Depression often occurs in the presence of one or more other disorders. For example, depression is reported to be at a higher rate in people with chronic obstructive pulmonary disease (COPD) than in the general population. COPD is a disease in which the lungs are damaged, making it difficult to breathe. Symptoms most commonly include chronic coughing and shortness of breath. A primary cause of COPD is cigarette smoking. Following a prescribed treatment plan is important for managing COPD. Unfortunately, people with COPD often do not adhere to their treatment plans. Being depressed makes adherence even more difficult. This study will evaluate the effectiveness of problem-solving therapy integrated with adherence-enhanced procedures (PSA) in treating older people with major depression and COPD.

Participants in this open label study will be randomly assigned to one of two groups: PSA or PID-C. In PSA, a therapist will teach participants problem-solving strategies focusing on treatment adherence, depressive symptoms, and disability. Participants will learn behaviors and solutions to help cope with these problems. In PID-C, a therapist will teach participants to identify obstacles to treatment adherence and to discover ways to overcome them. The treatment sessions for both groups will be initiated at the inpatient Pulmonary Unit of Burke Rehabilitation Hospital and will continue in the participants' homes. All participants will receive two treatment sessions during hospitalization, eight weekly sessions following discharge, and four monthly sessions after that. While hospitalized at Burke, participants will also undergo an assessment interview for 1.5 hours and another interview for 20 minutes 2 weeks following the initial assessment. Interviews lasting 1.5 hours will also occur in the homes of the participants at Weeks 10, 14, and 26 after discharge from Burke. All assessments will focus on depression severity, level of general functioning, and COPD treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Meets American Thoracic Society criteria for COPD
* Meets DSM-IV criteria for unipolar major depression
* Scores greater than 19 on 24-item Hamilton Depression Rating Scale
* Fluency in English sufficient for comprehending the questionnaires of the study and for understanding the therapists

Exclusion Criteria:

* Unable to give informed consent
* Experiencing suicidal thoughts
* History of or currently meets DSM-IV criteria for the following Axis I disorders: psychotic depression, psychotic disorder, bipolar disorder, dysthymic disorder, obsessive compulsive disorder, or current substance abuse
* Meets DSM-IV criteria for Axis II diagnosis of antisocial personality (by SCID-P and DSM-IV)
* Scores less than 24 on Mini-Mental State Exam (MMSE) or meets DSM-IV criteria for dementia
* Certain illnesses (e.g., untreated thyroid or adrenal disease, pancreatic cancer, lymphoma)
* Taking drugs known to cause depression (e.g., reserpine, alpha-methyl-dopa, steroids)
* Current involvement in psychotherapy
* Requires nursing home placement after discharge

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Measured at week 26

CONTACTS AND LOCATIONS:
Overall Officials: George S. Alexopoulos, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - The Burke Rehabilitation Hospital, White Plains, New York
  - Weill Medical College of Cornell University, White Plains, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Solomonov N, Kerchner D, Bein O, Lee CE, Diaz JL, Ciarleglio A, Kim S, Sirey JA, Gunning FM, Raue PJ, Banerjee S, Arean PA, Alexopoulos GS. Precision Assignment to Psychosocial Interventions for Late-Life Depression: An Automated Treatment Decision Rule. JAMA Psychiatry. 2025 Nov 1;82(11):1075-1084. doi: 10.1001/jamapsychiatry.2025.2518. PMID 40960814